CLINICAL TRIAL: NCT01172080
Title: Utility Analysis of an Endoscopy Follow-up System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Leffler, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010P000113
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Colonoscopy Adherence
Keywords: colonoscopy; adherence; reminders; quality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): Participants in this group are monitored for adherence to colonoscopy recommendations.
- intervention (Experimental): Participants to receive a protocol of reminder letters and a phone call regarding due follow up colonoscopy
  Interventions: Other: protocol of reminders regarding due colonoscopy

INTERVENTIONS:
Other: protocol of reminders regarding due colonoscopy — Participants receive two standardized letters followed by a phone call if they have not scheduled or completed their upcoming due colonoscopy
  Arms: intervention

SUMMARY:
Although systems are in place to ensure results of tests are communicated to patients, there is currently no generalized accepted strategy to ensure that patients undergo recommended follow-up testing. When follow-up tests are recommended months to years into the future, there is a high likelihood that the test will either be delayed or not performed resulting in the potential for poor outcomes and litigation. For this reason, there is a clear need for systems to be developed which automatically trigger patient communication when the date of a recommended follow-up test is approaching. The investigators propose to design a protocol for ensuring that patients are reminded to schedule follow-up tests and that this communication is documented in the online medical record. This work will provide the foundation for the creation of systems that significantly improve patient care, and can be easily adapted for use in many clinical departments and institutions.

Aim 1. To use patient focus groups to help design a system for improving adherence to endoscopy follow up recommendations

Aim 2. To develop a prototype endoscopy follow up system and test the effectiveness of the system on a cohort of patients due for a surveillance colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* due for a repeat surveillance colonoscopy for follow up of polyps during the study time period

Exclusion Criteria:

* not due for a repeat surveillance colonoscopy for follow up of polyps during the study time period

Max Age: 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 830 (Actual)
Dates: Start 2009-01; Primary Completion 2010-04 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
percentage of individuals scheduling colonoscopy | within three months of due date

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Leffler DA, Neeman N, Rabb JM, Shin JY, Landon BE, Pallav K, Falchuk ZM, Aronson MD. An alerting system improves adherence to follow-up recommendations from colonoscopy examinations. Gastroenterology. 2011 Apr;140(4):1166-1173.e1-3. doi: 10.1053/j.gastro.2011.01.003. Epub 2011 Jan 13. PMID 21237167